Association of Acupuncture and Cupping in Advanced Knee Osteoarthritis NCT 04168593

## Study protocol

120 patients waiting for surgical treatment from the knee outpatient clinic of the IOT-HCFMUSP were invited to participate in the project. Inclusion and exclusion criteria were applied, and those who accepted signed an informed consent form (ICF), and later allocated to the existing groups: A. Group A – Acupuncture Sham + Cupping Sham; B. Group B - Acupuncture Sham+ True Cupping; C. Group C - True Acupuncture + Cupping Sham; D. Group D – True Acupuncture + True Cupping. The Western Ontario and McMaster Osteoarthritis Index (WOMAC) questionnaire was used, which assesses pain, stiffness and functionality, and the number of analgesics and/or anti-inflammatory drugs used during the research period was also recorded. All the records were collected on the first interview and after 5 weeks treatment.

## Group A – Acupuncture Sham + Cupping Sham

Sham acupuncture: Placement of placebo "dagger" needles. The needle tip, when touching the patient's skin, retracts into itself without puncturing the skin. Application locations: LI11, SP9, SP10, LR8, GB34, ST34, Ex-LE5. Running time of 20 minutes. Sham cupping: after each acupuncture session (Sham or True), the respective needles were removed, and acrylic suction cups were placed over the region where the needles were, attached to a strip (micropore) without exerting any negative pressure or movement. Application time of 10 minutes.

Group B – Acupuncture Sham+ True Cupping Sham Acupuncture 20 min follow by 10 min of cupping around the knee

Group C – True Acupuncture + Cupping Sham 20 min of Acupuncture section follow by 10 min of Sham cupping around the knee

Group D – True Acupuncture + True Cupping 20 min of Acupuncture section follow by 10 min of cupping around the knee